CLINICAL TRIAL: NCT06700980
Title: Options for Lowering the Threshold to Brussels Out-of-hours Primary Care Services for Dutch Speaking Citizens
Acronym: BruWNed
Status: Recruiting | Type: Observational
Sponsor: Universitair Ziekenhuis Brussel (Other)
Collaborators: Brusselse Huisartsenkring (BHAK) (Unknown); Vlaamse Gemeenschapscommissie (VGC) (Unknown)
Responsible Party: Sponsor
Other Study IDs: 24366_BruWNed
Record Dates: First submitted 2024-11-07; First posted 2024-11-22 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Communication Barriers; Language; Primary Health Care; After-hours Care; Health Services Accessibility
Keywords: Language barrier; translation; healthcare; technological tool; Official language minority
MeSH Terms: conditions — Language | interventions — Focus Groups

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Focus Group: Four groups of participants will meet for online focus groups, identifying barriers and facilitators to the use of technological translation tools in Brussels out-of-hours primary care services for Dutch-speaking patients and French-speaking general practitioners.
  Interventions: Other: Focus Group

INTERVENTIONS:
Other: Focus Group — Dutch-speaking patients, Dutch- and/or French-speaking general practitioners and Dutch- and/or French-speaking representatives from pertinent organizational and policy sectors will be questioned in heterogeneous focus groups, identifying barriers and facilitators to the use of technological translation tools in Brussels out-of-hours primary care services for Dutch-speaking patients and French-speaking general practitioners.

SUMMARY:
The purpose of this qualitative study is to find out which technological translation tools can be used to improve Dutch-speaking care in all Brussels out-of-hours primary care services.

DETAILED DESCRIPTION:
Previous studies have shown that language barriers in healthcare can lead to communication problems between healthcare provider and patient. This can lead to a decrease in satisfaction, quality of care and patient safety. Dutch speakers are a minority in Brussels (a Dutch-French bilingual region in Belgium), and the majority of general practitioners (GPs) in the Brussels out-of-hours primary care services are French-speaking. Measures are already being taken to increase the number of bilingual (Dutch and French) GPs.

In addition, several technological tools (e.g. video interpreting, translation apps, ...) exist to overcome language barriers. The investigators want to explore which of these options can be used in Brussels out-of-hours primary care services to improve access for Dutch-speaking citizens. The objective of this study is to examine both barriers and facilitators to use these technological translation tools during language-discordant consultations with a French-speaking GP and a Dutch-speaking patient in Brussels out-of-hours primary care services.

To achieve this objective, the investigators aim to engage Dutch-speaking patients, Dutch- and/or French-speaking GPs, as well as Dutch- and/or French-speaking representatives from pertinent organizational and policy sectors.

There will be about 40 participants in total. Participants will answer questions during an online group session (focus group). There will be 4 focus groups, with a maximum of 10 participants in each focus group. Each focus group will last 60-90 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Patients: adult, living in Brussels, Dutch-speaking
* GPs: adult, working in Brussels, Dutch- and/or French-speaking
* Employees of professional organization-regulatory bodies: adult, Dutch-and/or French-speaking

Exclusion Criteria:

* Subject is not capable of will
* Subject cannot express themself in Dutch or French

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Dutch-speaking residents of Brussels Primary care physicians of Brussels Representatives from pertinent organizational and policy sectors of Belgium
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-12-10 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Exploration of barriers and facilitators of different stakeholders to the use of technological translation tools in Brussels out-of-hours primary care services for Dutch-speaking patients and French-speaking general practitioners. | The outcome will be measured during the online focus group, which will have a duration of 60 to 90 minutes.
  Focus group results will provide a list of barriers and facilitators to the use of technological translation tools in Brussels out-of-hours primary care services for Dutch-speaking patients and French-speaking general practitioners.

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Dr. A. Roex, Principal Investigator — Vrije Universiteit Brussel
Locations (1):
- Vrije Universiteit Brussel, Jette, Brussels Capital, Belgium

IPD SHARING:
Plan to Share IPD: No